CLINICAL TRIAL: NCT05600296
Title: Ultrasound-guided Ilioinguinal/Iliohypogastric Nerve Block Compared to the Combined Therapy With Spermatic Cord Block in Inguinal Herniotomy Operation in Children: a Randomized Controlled Study
Brief Title: Ultrasound-guided Ilioinguinal/Iliohypogastric Nerve Block Compared to the Combined Therapy With Spermatic Cord Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mona Gad 2
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Hernia, Inguinal
Keywords: inguinal herniotomy; ilioinguinal nerve block; iliohypogastric nerve block; spermatic cord block
MeSH Terms: conditions — Hernia, Inguinal | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ilioinguinal/iliohypogastric nerve block (IINB) (Active Comparator): evaluate the postoperative analgesic effects with using ultrasound-guided ilioinguinal/iliohypogastric nerve block (IINB) in children scheduled for elective open inguinal herniotomy.
  Interventions: Drug: Levobupivacaine; Procedure: Ilioinguinal/iliohypogastric nerve block (IINB)
- IINB+ Spermatic cord block (Active Comparator): evaluate the postoperative analgesic effects with using ultrasound-guided IINB + spermatic cord block (SCB) in children scheduled for elective open inguinal herniotomy.
  Interventions: Drug: Levobupivacaine; Procedure: IINB+ Spermatic cord block

INTERVENTIONS:
Drug: Levobupivacaine — Evaluation the postoperative analgesic effects by using ultrasound-guided spermatic cord block (SCB) and IINB in children scheduled for elective open inguinal herniotomy. The study hypothesized that, the combined block with SCB and IINB would result in more effective postoperative analgesia than the use of IINB alone.
Procedure: Ilioinguinal/iliohypogastric nerve block (IINB) — Ilioinguinal/iliohypogastric nerve block (IINB)
  Arms: Ilioinguinal/iliohypogastric nerve block (IINB)
Procedure: IINB+ Spermatic cord block — IINB+ Spermatic cord block
  Arms: IINB+ Spermatic cord block

SUMMARY:
This is a single center randomized, controlled, double-blinded, noninferiority study. Male pediatric patients who underwent inguinal herniotomy will be screened for eligibility. Patients will be randomly allocated to IINB and IINB/SCB groups with allocation ratio 1:1. The primary outcome measure will be the proportion of patients who needed rescue analgesia during the first postoperative 6 h. The secondary outcome measures will be intraoperative heart rate and mean arterial blood pressure (MAP), the postoperative pain FLACC pain scale, and intravenous paracetamol consumption, the incidence of adverse effects including hematoma, postoperative vomiting and fever.

DETAILED DESCRIPTION:
Inguinal herniotomy in children is a frequent surgical procedure that require good postoperative analgesia. Ultrasound-guided ilioinguinal/iliohypogastric nerve block is a widely validated anesthetic technique for this procedureز

Currently, central neuraxial analgesic techniques have been replaced by ultrasoundguided interfascial plane blocks that have gained more popularity among anesthetists because they are safer, easily performed, associated with minor hemodynamic changes and can be done in the presence of contraindications of the neuraxial block .

Ultrasound-guided ilioinguinal/iliohypogastric nerve block (IINB) is commonly done in pediatric patients to control pain after lower abdominal surgeries and has been shown to be effective in controlling pain after inguinal hernia repair .

However IINB don't affect the genitofemoral neve that contributes the sensory innervation of the inguinal region. The spermatic cord (SC) is a unique male structure that contains the vas deferens, testicular arteries, the pampiniform plexus of veins, and the ilioinguinal nerve and genital branch of the genitofemoral nerve (GFN). To provide complete analgesia for inguinal hernia surgery, GFN should be blocked in addition to IINB .

ELIGIBILITY:
Inclusion Criteria:

* Male pediatric patients
* underwent elective open unilateral inguinal herniotomy
* Informed written consent will be obtained from the parents or the legal guardian.

Exclusion Criteria:

* local infection at the puncture site,
* bleeding disorder,
* allergy to amide local anesthetics,
* history of clinically significant cardiac, hepatic, or renal disorders.
* neurological dysfunction

Ages: 12 Months to 60 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Rescue Analgesia | From base line to 6 hours postoperatively
  Assessment of the proportion of patients who needed rescue analgesia. Intravenous paracetamol 15mg/kg will be given as a rescue analgesic if FLACC pain scale ≥ 4
Post Operative Pain | From base line to 6 hours postoperatively
  Assessment of The pain level of the cases by (Face, Leg, Activity, Cry, Consolability) pain scale (FLACC ) means of the digital pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Gad, Assist.Prof., Principal Investigator — Department of anesthesia and SICU,Faculty of medicine,Mansoura university , Egypt.
Locations (1):
- Mansoura university Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No